CLINICAL TRIAL: NCT02455141
Title: Epirubicin-Cyclophosphamide Followed by Taxanes or Taxanes Plus Carboplatin in Triple-Negative Breast Cancer：A Prospective, Randomized, Phase III Trial
Brief Title: Adjuvant Treatment of EC Followed by Taxane +/- Carboplatin in Triple-Negative Breast Cancer
Acronym: TCTN
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Kunwei Shen, professor, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RJBC1501
Record Dates: First submitted 2015-05-02; First posted 2015-05-27 (Estimated); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Breast Neoplasm
Keywords: chemptherapy; triple negative; taxanes; carboplatin
MeSH Terms: conditions — Breast Neoplasms | interventions — Epirubicin; Cyclophosphamide; Taxoids; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Taxanes (Active Comparator): Epirubicin plus Cyclophosphamide followed by Paclitaxel or Docetaxel
  Interventions: Drug: Epirubicin plus Cyclophosphamide; Drug: Taxanes
- Taxanes plus carboplatin (Experimental): Epirubicin plus Cyclophosphamide followed by Paclitaxel or Docetaxel + Carboplatin
  Interventions: Drug: Epirubicin plus Cyclophosphamide; Drug: Taxanes plus Carboplatin

INTERVENTIONS:
Drug: Epirubicin plus Cyclophosphamide — Epirubicin 90mg/m2, d1, q3w*4 Cyclophosphamide: 600mg/m2, d1, q3w*4
  Other Names: EC
Drug: Taxanes — Paclitaxel: 80mg/m2, d1, qw*12 or Docetaxel: 80-100mg/m2,d1,q3w*4
  Arms: Taxanes
Drug: Taxanes plus Carboplatin — Paclitaxel: 80mg/m2, d1,d8,d15, q4w*4 Carboplatin AUC=2, d1,d8,d15, q4w*4 or Docetaxel: 75mg/m2,d1,q3w*4 plus Carboplatin AUC=5-6, d1, q3w*4
  Arms: Taxanes plus carboplatin

SUMMARY:
To compare disease-free survival (DFS) rate of adjuvant chemotherapy epirubicin-cyclophosphamide followed by weekly paclitaxel or docetaxel (EC-T), or weekly paclitaxel or docetaxel-carboplatin (EC-TCb) in triple-negative breast cancer.

DETAILED DESCRIPTION:
This study plans to enroll triple-negative breast cancer patients who have complete tumor removal. Patients are randomized to receive either EC-wP/T or EC-wP/TCb adjuvant chemotherapy. For triple-negative breast cancer, a subgroup of triple-negative breast cancer has DNA repairement deficiency and adding carboplatin to paclitaxel may improve DFS on the basis of weekly paclitaxel adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria

* Histologically confirmed adenocarcinoma of the breast, completely tumor removal by either modified radical mastectomy or local excision plus axillary lymph node dissection (i.e., breast conservation therapy) or sentinel node biopsy. (Tumor-free margins at least 1 mm for both invasive and noninvasive carcinoma except for lobular carcinoma in situ (less than 1 mm allowed);
* Tumor specimens are available for estrogen receptor (ER), progesterone receptor (PgR) and Her2 (human epidermal-growth-factor receptor 2) detection, patients should be with triple negative breast cancer. Triple-negative disease is defined as ER <10% positivity, PgR <10% positivity, and negativity for Her2 (IHC (immunohistochemistry) 0-1+ or FISH (fluorescence in situ hybridization) negative);
* Adequate bone marrow function
* Adequate liver and renal function
* Eastern Cooperative Oncology Group (ECOG) Performance Score 0-1;
* Women with potential child-bearing must have a negative pregnancy test (urine or serum) within 7 days of drug administration and agree to use an acceptable method of birth control to avoid pregnancy for the duration of the study;
* Written informed consent according to the local ethics committee requirements.

Exclusion Criteria:

* Prior systemic of breast cancer, including chemotherapy;
* Metastatic breast cancer;
* With a history of malignant tumor except uterine cervix cancer in situ or skin basal cell carcinoma;
* Patients with medical conditions that indicate intolerant to adjuvant therapy and related treatment, including uncontrolled pulmonary disease, diabetes mellitus, severe infection, active peptic ulcer, coagulation disorder, connective tissue disease or myelo-suppressive disease;
* Has active hepatitis B or hepatitis C with abnormal liver function tests (LFTs) or is known to be HIV positive;
* Contraindication for using dexamethasone;
* History of congestive heart failure, uncontrolled or symptomatic angina pectoris, arrhythmia or myocardial infarction; poorly controlled hypertension (systolic BP>180 mmHg or diastolic BP>100 mmHg);
* Has peripheral neuropathy no less than grade 1;
* Patient is pregnant or breast feeding;
* Patients with psychiatric disorder or other diseases leading to incompliance to the therapy;
* Known severe hypersensitivity to any drugs in this study;
* Treatment with any investigational drugs within 30 days before the beginning of study treatment.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 786 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | From time of randomization to 5 years after enrollment.
  The time from randomization to local or regional recurrence, distant metastases, other non-breast secondary primary malignancies, contralateral breast cancer, or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Distant disease-free survival | From time of randomization to 5 years after enrollment.
  The time from randomization to distant metastases, other non-breast secondary primary malignancies, or death due to any cause, whichever occurs first.
Overall Survival | From time of randomization to 5 years after enrollment.
  The time from randomization to death due to any cause.
Incidence of adverse events | From randomization to four weeks after end of study treatment
  To compare the grade 3-5 adverse events among two treatment arms according to the NCI-CTCAE v4.0 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Kunwei Shen, professor, Principal Investigator — Affiliated Ruijin Hospital of Shanghai JiaoTong University School of Medicine
Locations (27):
- China (27):
  - Fuding Hospital, Fuding, Fujian
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Quanzhou First Hospital, Quanzhou, Fujian
  - Foshan No.1 People's Hospital, Foshan, Guangdong
  - Guangdong Maternal and Child Health Care Hospital, Guangzhou, Guangdong
  - Cancer Hospital Affiliated to Harbin Medical University, Harbin, Heilongjiang
  - Jiangsu Jiangyin People's Hospital, Jiangyin, Jiangsu
  - The First People's Hospital of Wujiang District, Suzhou, Jiangsu
  - Yancheng Hospital of TCM, Yancheng, Jiangsu
  - Obstetrics & Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanghai JiaoTong University School of Medicine, Ruijin Hospital, Shanghai, Shanghai Municipality
  - Central Hospital of Huangpu District, Shanghai, Shanghai, Shanghai Municipality
  - Shanghai International Peace Maternal and child health care hospital, Shanghai, Shanghai Municipality
  - The Ninth People's Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Hangzhou Cancer Hospital, Hangzhou, Zhejiang
  - Zhejiang Provincial Hospital of TCM, Hangzhou, Zhejiang
  - Jiaxin Maternal and Child Health Care Hospital, Jiaxin, Zhejiang
  - Lishui People's Hospital, Lishui, Zhejiang
  - Ningbo Medical Treatment Center Lihuili Hospital, Ningbo, Zhejiang
  - Ningbo Women and Children's Hospital, Ningbo, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
  - Rui'an People's Hospital, Rui’an, Zhejiang
  - Shaoxing Shangyu People's Hospital, Shaoxing, Zhejiang
  - Shaoxing No.2 Hospital, Shaoxing, Zhejiang
  - Taizhou Central Hospital, Taizhou, Zhejiang
  - Wenzhou People's Hospital, Wenzhou, Zhejiang
  - Zhoushan Hospital, Zhoushan, Zhejiang

REFERENCES:
- [Background] Hayes DF, Thor AD, Dressler LG, Weaver D, Edgerton S, Cowan D, Broadwater G, Goldstein LJ, Martino S, Ingle JN, Henderson IC, Norton L, Winer EP, Hudis CA, Ellis MJ, Berry DA; Cancer and Leukemia Group B (CALGB) Investigators. HER2 and response to paclitaxel in node-positive breast cancer. N Engl J Med. 2007 Oct 11;357(15):1496-506. doi: 10.1056/NEJMoa071167. PMID 17928597
- [Background] Martin M, Rodriguez-Lescure A, Ruiz A, Alba E, Calvo L, Ruiz-Borrego M, Santaballa A, Rodriguez CA, Crespo C, Abad M, Dominguez S, Florian J, Llorca C, Mendez M, Godes M, Cubedo R, Murias A, Batista N, Garcia MJ, Caballero R, de Alava E. Molecular predictors of efficacy of adjuvant weekly paclitaxel in early breast cancer. Breast Cancer Res Treat. 2010 Aug;123(1):149-57. doi: 10.1007/s10549-009-0663-z. PMID 20037779
- [Background] Sikov WM, Berry DA, Perou CM, Singh B, Cirrincione CT, Tolaney SM, Kuzma CS, Pluard TJ, Somlo G, Port ER, Golshan M, Bellon JR, Collyar D, Hahn OM, Carey LA, Hudis CA, Winer EP. Impact of the addition of carboplatin and/or bevacizumab to neoadjuvant once-per-week paclitaxel followed by dose-dense doxorubicin and cyclophosphamide on pathologic complete response rates in stage II to III triple-negative breast cancer: CALGB 40603 (Alliance). J Clin Oncol. 2015 Jan 1;33(1):13-21. doi: 10.1200/JCO.2014.57.0572. Epub 2014 Aug 4. PMID 25092775
- [Background] von Minckwitz G, Schneeweiss A, Loibl S, Salat C, Denkert C, Rezai M, Blohmer JU, Jackisch C, Paepke S, Gerber B, Zahm DM, Kummel S, Eidtmann H, Klare P, Huober J, Costa S, Tesch H, Hanusch C, Hilfrich J, Khandan F, Fasching PA, Sinn BV, Engels K, Mehta K, Nekljudova V, Untch M. Neoadjuvant carboplatin in patients with triple-negative and HER2-positive early breast cancer (GeparSixto; GBG 66): a randomised phase 2 trial. Lancet Oncol. 2014 Jun;15(7):747-56. doi: 10.1016/S1470-2045(14)70160-3. Epub 2014 Apr 30. PMID 24794243
- [Background] Chen XS, Yuan Y, Garfield DH, Wu JY, Huang O, Shen KW. Both carboplatin and bevacizumab improve pathological complete remission rate in neoadjuvant treatment of triple negative breast cancer: a meta-analysis. PLoS One. 2014 Sep 23;9(9):e108405. doi: 10.1371/journal.pone.0108405. eCollection 2014. PMID 25247558
- [Derived] Chen X, Huang J, Shi H, Zhu J, Wu W, Ye G, He Q, Shi Y, Zhang A, Xie X, Wang X, Chen X, Wu W, Wu J, Li Z, Li Z, Dai Y, Ren W, Shao Q, Chen Y, Zeng Y, Zhang F, Dong S, Pegram MD, Shen K. Adjuvant Epirubicin Plus Cyclophosphamide Followed by Taxanes With or Without Carboplatin in Early-Stage Triple-Negative Breast Cancer (RJBC 1501): A Randomized Phase III Trial. J Clin Oncol. 2026 Jan 20;44(3):143-152. doi: 10.1200/JCO-25-02412. Epub 2025 Dec 9. PMID 41365333